CLINICAL TRIAL: NCT06002503
Title: A Phase I, Randomized, Observer-Blind Trial to Assess the Safety, Reactogenicity and Immunogenicity of a Venezuelan Equine Encephalitis (VEE) DNA Vaccine Candidate Administered Intramuscularly and Intradermally by Jet Injection to Healthy Adults
Brief Title: Safety, Reactogenicity and Immunogenicity of a Venezuelan Equine Encephalitis DNA Vaccine Candidate Administered by Jet Injection
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaJet, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VEEV-PJ-01
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-03

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- 1: Intramuscular (Experimental): Route (device): Intramuscular (PharmaJet Stratis Needle-free Injection System) Vaccine dose schedule (week): 0, 4, 8 Saline dose schedule (week): 26
  Interventions: Drug: Venezuelan Equine Encephalitis DNA Vaccine; Device: PharmaJet Stratis Needle-free Injection System
- 2: Intramuscular (Experimental): Route (device): Intramuscular (PharmaJet Stratis Needle-free Injection System) Vaccine dose schedule (week): 0, 8, 26 Saline dose schedule (week): 4
  Interventions: Drug: Venezuelan Equine Encephalitis DNA Vaccine; Device: PharmaJet Stratis Needle-free Injection System
- 3: Intradermal (Experimental): Route (device): Intradermal (PharmaJet Tropis Needle-free Injection System) Vaccine dose schedule (week): 0, 4, 8 Saline dose schedule (week): 26
  Interventions: Drug: Venezuelan Equine Encephalitis DNA Vaccine; Device: PharmaJet Tropis Needle-free Injection System
- 4: Intradermal (Experimental): Route (device): Intradermal (PharmaJet Tropis Needle-free Injection System) Vaccine dose schedule (week): 0, 8, 26 Saline dose schedule (week): 4
  Interventions: Drug: Venezuelan Equine Encephalitis DNA Vaccine; Device: PharmaJet Tropis Needle-free Injection System

INTERVENTIONS:
Drug: Venezuelan Equine Encephalitis DNA Vaccine — Venezuelan Equine Encephalitis DNA Vaccine Candidate
Device: PharmaJet Stratis Needle-free Injection System — Intramuscular Needle-free Injection System (Jet Injector)
  Arms: 1: Intramuscular; 2: Intramuscular
Device: PharmaJet Tropis Needle-free Injection System — Intradermal Needle-free Injection System (Jet Injector)
  Arms: 3: Intradermal; 4: Intradermal

SUMMARY:
The goal of this clinical trial is to evaluate the safety and reactogenicity of a VEE DNA Vaccine candidate delivered by either intramuscular or intradermal jet injection. The main question it aims to answer is:

• Is the VEE DNA Vaccine candidate safe

Participants will:

* Receive the VEE DNA Vaccine candidate by either intramuscular or intradermal jet injection
* Provide blood and urine samples
* Complete ECGs
* Complete physical exams
* Complete diaries

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, male or female.
* Ages at least 18 at the start of the study and no greater than 49 years of age on Day 1 of vaccination.
* Participants must be available for all visits and for the complete duration of the study.
* Participants must, in the opinion of the Investigator or person obtaining consent, understand the information provided and be capable of providing informed consent.
* Women of child bearing potential (WOCBP) must have a negative pregnancy test and be willing to use an effective method of contraception: oral contraception, diaphragm, cervical cap, intrauterine device, condom, or be anatomically sterile (in self or partner) from the date of screening until at least 6 months after the last vaccination.
* If subject is a sexually active male, must be willing to use an effective method of contraception (such as condoms or be anatomically sterile) from screening until 6 months after the last vaccination.

Exclusion Criteria:

* Clinically relevant abnormality on history or examination including a history of immunodeficiency or use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered to be significant by the designated trial physician in the last 6 months.
* Any acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that, in the opinion of the Investigator, would preclude participation.
* Any of the following laboratory parameters with abnormal values that are moderate in severity: hematology (hemoglobin, absolute neutrophil count, absolute lymphocyte count, platelets); urinalysis; biochemistries (total bilirubin, creatinine, AST, ALT).
* If female, pregnant, lactating, or planning pregnancy within 6 months of the final vaccination.
* Receipt of a blood transfusion or blood products 6 months prior to enrollment.
* Participation in another clinical trial of an investigational product currently or within the past 12 weeks or expected participation during the study.
* History of severe local or systemic reactions to vaccination or a history of severe allergic reactions.
* History of Guillain-Barre syndrome.
* Confirmed diagnosis of HBV infection (surface antigen positive, HBsAg); Hepatitis C infection (HCV Ab positive); HIV infection, or active syphilis.
* History of grand mal epilepsy, or currently taking anti-epileptics.
* Any condition associated with prolonged bleeding time, which would contraindicate skin or muscle injection.
* Abnormal ECG finding that, in the opinion of the Investigator, excludes the subject from participating.
* History of syncope or history of a fainting episode within one year of study entry.
* Extensive tattoos or markings covering the eligible sites of administration (the skin or muscle of the upper left and right deltoid muscles).
* Presence of any surgical/traumatic metal implants, or significant scar tissue that may impair appropriate injection at the eligible sites of administration (skin or muscle of the upper left and right deltoid muscles).
* In the opinion of the Investigator, is unlikely to comply with the protocol.
* As confirmed/reported by the study subject, a history of: exposure to Venezuelan Equine Encephalitis Virus (VEEV) or related alphavirus; prior immunization with an alphavirus replicon-based vaccine; prior immunization with a live-attenuated alphavirus vaccine; prior immunization with an inactivated alphavirus vaccine.
* A history of encephalitis as confirmed/reported by the study subject.
* Prior immunization against VEEV or related alphavirus or encephalitis, as confirmed/reported by the study subject.
* History of alcohol abuse, illicit drug use, physical dependence on any opioid, or any history of drug abuse (excluding marijuana) or addiction within 12 months of screening.
* Involved in the planning or conduct of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with immediate reactions | 30 minutes after each vaccination
  The nature, frequency, and severity of immediate reactions following vaccination
Solicited adverse events | 7 days after each vaccination
  The nature, frequency, and severity of solicited adverse events
Unsolicited adverse events | 28 days after the final vaccination
  The nature, frequency, and severity of unsolicited adverse events
Adverse events | 1 year
  The nature, frequency, and severity of adverse events

SECONDARY OUTCOMES:
VEEV-specific antibody | 1 year
  PsVNA50
Seroconversion rate | 1 year
  PsVNA50

CONTACTS AND LOCATIONS:
Locations (1):
- Velocity Clinical Research, Cincinnati, Ohio, United States